CLINICAL TRIAL: NCT03381404
Title: An Open-label, Mass Balance Study to Investigate the Absorption, Metabolism and Excretion of [14C]-MT-8554 After a Single Oral Dose to Healthy Male Subjects
Brief Title: Mass Balance Study With MT-8554
Acronym: MT-8554 MB
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MT-8554-E07; 2017-002830-21 (EudraCT Number)
Record Dates: First submitted 2017-11-29; First posted 2017-12-22 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteer
Keywords: Mass Balance Study with MT-8554

STUDY DESIGN:
Intervention Model Description: Open Label
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- [14C] MT-8554 (Experimental)
  Interventions: Drug: [14C] MT-8554

INTERVENTIONS:
Drug: [14C] MT-8554 — 14-C MT-8554

SUMMARY:
This is a single-centre, open-label, mass balance study in healthy male subjects utilising a single oral dose of [14C] MT 8554.

ELIGIBILITY:
Inclusion Criteria:

* 1. Able to provide written informed consent to participate in this study after reading the participant information sheet and informed consent form and after having the opportunity to discuss the study with the Investigator or designee.
* 2. Healthy and free from clinically significant illness or disease as determined by medical history, physical examination, laboratory and other tests at Screening and Day 1.
* 3. Male Caucasian subjects, aged 30 to 55 years (inclusive) at Screening.
* 4. A body weight of ≥60 kg and a body mass index (Quetelet index) ranging from 18 to 30 kg/m2 (inclusive) at Screening or Day 1.
* 5. Subjects and partners agree to use contraception throughout the study as detailed in the Protocol body.
* 6. In the Investigator's opinion, subject is able to understand the nature of the study and any risks involved in participation, and willing to cooperate and comply with the Protocol restrictions and requirements.
* 7. Regular daily bowel movements (i.e., production of at least one stool per day).

Exclusion Criteria:

* 1. Previously having received MT-8554.
* 2. Participation in more than three clinical studies involving administration of an IMP in the previous year, or any study within 12 weeks (or, if relevant, five half-lives, whichever is the longer) prior to dosing.
* 3. Presence or history of severe adverse reaction or allergy to any medicinal product that is of clinical significance.
* 4. Subjects who have received any prescribed systemic or topical medication within 14 days (or, if relevant, five half-lives, whichever is longer) prior to dosing unless, in the opinion of the Investigator and Sponsor, the medication will not interfere with the study procedures or compromise safety. Subjects who have received slow release medicinal formulations considered to still be active within 14 days (or, if relevant, five half-lives, whichever is longer) prior to dosing will also be excluded unless, in the opinion of the Investigator or Sponsor, the medication will not interfere with the study procedures or compromise subject safety.
* 5. Subjects who have used any non-prescribed systemic or topical medication (including herbal remedies) within 7 days (or, if relevant, five half-lives, whichever is longer) prior to dosing unless, in the opinion of the Investigator and Sponsor, the medication will not interfere with the study procedures or compromise subject safety. Occasional use (2 g/day for 3 days) of paracetamol (acetaminophen) for mild analgesia is permitted.
* 6. Subjects who have received any medications, including St John's Wort, known to chronically alter drug absorption or elimination processes within 30 days (or, if relevant, five half-lives, whichever is longer) prior to dosing unless, in the opinion of the Investigator and Sponsor, the medication will not interfere with the study procedures or compromise subject safety.
* 7. Clinically significant (in the opinion of the Investigator) endocrine, thyroid, hepatic (including Gilbert's syndrome), respiratory, gastrointestinal, renal, cardiovascular disease or history (within the last 2 years) of any significant psychiatric/psychotic illness disorder (including anxiety, depression and reactive depression).
* 8. Clinically relevant abnormal medical history, physical findings or laboratory values at Screening or Day 1 that could interfere with the objectives of the study or compromise subject safety, as judged by the Investigator.
* 9. Subjects with aspartate aminotransferase, alanine aminotransferase ≥1.5 × upper limit of normal or total bilirubin or creatine kinase above the reference range at Screening or Day 1.
* 10. Subjects with creatinine clearance <60 mL/min (calculated using the Cockcroft-Gault-formula) at Screening.
* 11. Family history of long or short QT syndrome, syncope of unknown cause or Torsades de Pointes.
* 12. Clinically significant 12-lead electrocardiogram (ECG) abnormalities, including subjects with corrected QT interval using Fridericia's formula (QTcF) of >450 ms, at Screening or Day 1, confirmed by repeat assessment.
* 13. Blood pressure (supine) at Screening or Day 1 outside the range of 90 to 140 mmHg (systolic) or 50 to 90 mmHg (diastolic) and pulse rate outside the range of 40 to 100 beats per minute, confirmed by repeat assessment. Evidence of postural hypotension at Screening defined as a decrease of >20 mmHg in systolic or >10 mmHg in diastolic blood pressure between the supine and standing position, confirmed by repeat assessment.
* 14. Tympanic body temperature at Day 1 that is outside the local reference range (35.5°C to 37.8°C), confirmed by repeat assessment.
* 15. Excessive consumption of food or drink containing caffeine, including coffee, tea, cola, energy drinks or chocolates (≥5 cups of coffee or equivalent per day).
* 16. Presence or history of drug abuse (as defined by Diagnostic and Statistical Manual of Mental Disorders [DSM-V] criteria) or a positive urine test for drugs of abuse at Screening or Day 1.
* 17. Presence or history (in the last 2 years) of alcohol abuse, or intake of more than 28 units/224 g of alcohol weekly or a positive breath test for alcohol at Screening or Day 1. One unit/8 g is equivalent to a half-pint (280 mL) of beer or one measure (25 mL) of spirits or one glass (125 mL) of wine.
* 18. Subjects who use tobacco or nicotine-containing products (cigarettes, snuff, chewing tobacco, cigars, pipes, e cigarettes or nicotine-replacement products) within 3 months prior to dosing, or positive urine cotinine test at Screening or Day 1.
* 19. Test positive for hepatitis B surface antigen, hepatitis B core antibody, hepatitis C antibody or human immunodeficiency virus (HIV) 1 and HIV 2 antibodies at Screening.
* 20. Donate one or more units of blood (450 mL) within 3 months prior to Screening, or plasma within 7 days prior to Screening, or platelets within 6 weeks prior to Screening, or intention to donate blood within 3 months after the last scheduled visit.
* 21. Consumption of food or drink containing red wine, Seville oranges (including marmalade), liquorice, cranberry (including fruit juice) or grapefruit (including fruit juice) from 7 days prior to Day 1.
* 22. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs, or which may jeopardise the subject in case of participation in the study. The Investigator should be guided by evidence of any of the following:
* 23. History of irritable bowel syndrome, or other manifestation of abnormal bowel habit (e.g., diarrhoea, constipation);
* 24. History of inflammatory bowel disease, gastritis, ulcers, gastrointestinal or rectal bleeding;
* 25. History of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy or bowel resection;
* 26. History or clinical evidence of pancreatic injury or pancreatitis.
* 27. Radiation exposure, excluding background radiation but including that from the present study, diagnostic X-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 1999, shall participate in the study.

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2018-01-29 (Actual); Study Completion 2018-01-29 (Actual)

PRIMARY OUTCOMES:
Total radioactivity in urine and faeces | Up to 14 Days after dosing
Maximum observed plasma concentration [Cmax] | Up to 14 Days after dosing
Time at which Cmax occurs [tmax] | Up to 14 Days after dosing
Area under the plasma concentration-time curve from time zero to the last measurable concentration [AUC0-last] | Up to 14 Days after dosing
Apparent terminal elimination half-life [t1/2] | Up to 14 Days after dosing
Terminal elimination rate constant [Kel] | Up to 14 Days after dosing

SECONDARY OUTCOMES:
Safety and tolerability as measured by adverse events (AEs) | Up to 14 Days after dosing
Safety and tolerability as measured by vital signs | Up to 14 Days after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Head of Medical Science, Study Director — Tanabe Pharma America, Inc.
Locations (1):
- Investigational center, City Name, United Kingdom